CLINICAL TRIAL: NCT01358916
Title: Improvement of Antibiotic Prescription in Outpatient Care: a Cluster-randomised Intervention Study Using a Sentinel Surveillance Network of Physicians
Brief Title: Intervention Study to Improve Antibiotic Prescription in Outpatient Care
Acronym: SAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Bundesamt für Gesundheit (Unknown); Sentinella Netzwerk (Unknown); Schweizerische Gesellschaft für Infektiologie (Unknown); Pädiatrische Infektiologie Gruppe Schweiz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Swiss Federal Office of Health
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections
Keywords: antimicrobial resistance; antibiotic prescription; primary health care; cluster-randomized trial
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual information policy (No Intervention): No specific intervention
- Antibiotic therapy guidelines (Other)
  Interventions: Other: Mailing of antibiotic therapy guidelines to the sentinel physicians

INTERVENTIONS:
Other: Mailing of antibiotic therapy guidelines to the sentinel physicians — Mailing of antibiotic therapy guidelines to the sentinel physicians and regular feedback on antibiotic prescription
  Arms: Antibiotic therapy guidelines

SUMMARY:
Antimicrobial resistance has become a world-wide problem and antibiotic consumption is a major driving force for the development of resistance. Thus optimization of antibiotic prescription and reduction of unnecessary antimicrobial treatment are essential in the prevention and reduction of antimicrobial resistance rates.

The goal of this study is the improvement of antibiotic prescription in outpatient care. The study will take place within a Swiss-wide sentinel surveillance network of physicians. The participating physicians will be randomised in a control and intervention group. The intervention group will receive therapeutic guidelines for the treatment of upper and lower respiratory tract infections and lower urinary tract infection as well as regular feed-backs on the prescription pattern of the sentinel physicians during the past months. Sentinel physicians will collect information about each antibiotic prescription, its indication and characteristics of the patient.

Our hypothesis is that the prescription pattern in the intervention group will be optimised and unnecessary antibiotic therapy will be reduced compared to the control group.

DETAILED DESCRIPTION:
Background

Antimicrobial resistance has become a world-wide problem and antibiotic consumption is a major driving force for the development of resistance. Thus optimization of antibiotic prescription and reduction of unnecessary antimicrobial treatment are essential in the prevention and reduction of antimicrobial resistance rates.

The goal of this study is the qualitative and quantitative improvement of antibiotic prescription in outpatient care. The study will take place within a Swiss-wide sentinel surveillance network consisting of general practitioners, pediatricians and physicians specialized in internal medicine. The participating physicians will be randomised in a control and intervention group. The intervention group will receive therapeutic guidelines for the treatment of upper and lower respiratory tract infections and lower urinary tract infections. Furthermore, regular feed-backs on the prescription pattern of the sentinel physicians in the last months will be provided.

Information about each antibiotic prescription, its indication and the characteristics of the patients will be collected by the sentinel physicians. The standardized reporting of antibiotic prescription by sentinel physicians has been carried out in Switzerland since 2006.

Our hypothesis is that the intervention will affect the antibiotic prescription pattern and that the investigators will observe an optimization of antibiotic prescription and a decrease in the number of antibiotic prescriptions.

Objective

Primary goals:

* Increase of the percentage of penicillin prescriptions for upper and lower respiratory tract infections
* Increase of the percentage of TMP/SMX prescriptions for lower urinary tract infections in adults

Secondary goal:

* Decrease of the percentage of quinolone prescriptions for COPD exacerbations in adults
* Decrease of the number of antibiotic prescriptions for sinusitis and other upper respiratory tract infections

Methods

Prospective cluster-randomised intervention study. The intervention is the mailing of treatment guidelines for upper and lower respiratory tract infections and lower urinary tract infections as well as regular feed-backs on the antibiotic prescription patterns of the sentinel physicians during the past months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory tract infections or urinary tract infections

Exclusion Criteria

* Patients with chronic disease requiring regular antibiotic treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of prescriptions of penicillin for respiratory tract infections | Two years
Percentage of prescriptions of TMP/SMX for lower urinary tract infections in adults | Two years

SECONDARY OUTCOMES:
Percentage of prescriptions of quinolone for COPD exacerbations in adults | Two years
Percentage of antibiotic prescriptions for the indications "sinusitis" and "other upper respiratory tract infections" | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kronenberg, Dr. med., Principal Investigator — University of Bern
Locations (1):
- Institute for Infectious Diseases, Bern, Switzerland

REFERENCES:
- [Derived] Hurlimann D, Limacher A, Schabel M, Zanetti G, Berger C, Muhlemann K, Kronenberg A; Swiss Sentinel Working Group. Improvement of antibiotic prescription in outpatient care: a cluster-randomized intervention study using a sentinel surveillance network of physicians. J Antimicrob Chemother. 2015 Feb;70(2):602-8. doi: 10.1093/jac/dku394. Epub 2014 Oct 17. PMID 25326088